CLINICAL TRIAL: NCT06860529
Title: Serplulimab Combined With Chemotherapy for Early-stage HR+/HER2- Breast Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, Zhenzhen Liu, Professor, Henan Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HELEN-018plus
Record Dates: First submitted 2025-02-05; First posted 2025-03-06 (Actual); Last update posted 2025-06-23 (Actual); Status verified 2025-06

CONDITIONS: HR+/HER2- Breast Cancer
MeSH Terms: interventions — Epirubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental: Treatment group1 (Experimental): NabPE+Serplulimab group（Epirubicin ivgtt on Day 1+Albumin Paclitaxel ivgtt on Day 1+Serplulimab ivgtt on Day 3）
  Interventions: Drug: Serplulimab; Drug: Epirubicin; Drug: Albumin Paclitaxel
- Experimental: Treatment group2 (Experimental): NabPE+Serplulimab group（Epirubicin ivgtt on Day 1+Albumin Paclitaxel ivgtt on Day 1+Serplulimab ivgtt on Day 1）
  Interventions: Drug: Serplulimab; Drug: Epirubicin; Drug: Albumin Paclitaxel
- Control group (Active Comparator): NabPE(Epirubicin ivgtt on Day 1+Albumin Paclitaxel ivgtt on Day 1）
  Interventions: Drug: Epirubicin; Drug: Albumin Paclitaxel

INTERVENTIONS:
Drug: Serplulimab — Serplulimab is administered intravenously
  Arms: Experimental: Treatment group1; Experimental: Treatment group2
Drug: Epirubicin — Epirubicin ivgtt
Drug: Albumin Paclitaxel — Albumin Paclitaxel ivgtt

SUMMARY:
The neoadjuvant treatment options commonly used for HR+/HER2- breast cancer are mainly anthracycline sequential or combined with paclitaxel chemotherapy regimens. Several clinical studies have confirmed that albumin paclitaxel is more effective than solvent-based paclitaxel, and therefore, albumin paclitaxel in combination with epirubicin has also become a commonly used chemotherapy regimen in clinical practice.

The aim of this study was to explore the efficacy and safety of the Serplulimab combined with nab-paclitaxel and epirubicin in the neoadjuvant treatment of HR+/HER2- breast cancer

ELIGIBILITY:
3.1 Inclusion Criteria

Patients must meet all of the following criteria to be eligible:

Age: ≥18 years old.

Clinical-pathological confirmation:

cT2-cT4 breast cancer, or cT1c with axillary lymph node metastasis.

Histopathologically confirmed HR+/HER2- invasive breast cancer:

ER and/or PR positive (IHC nuclear staining ≥1%).

HER2-negative (IHC 0 or 1+ without FISH testing, or IHC 2+ with FISH-negative amplification).

Ki67 ≥20%.

Clinically measurable lesions:

Measurable lesions confirmed by ultrasound, mammography, or MRI (optional) within 1 month prior to randomization.

Adequate organ and bone marrow function (within 1 month prior to chemotherapy):

Absolute neutrophil count (ANC) ≥2.0 × 10^9/L.

Hemoglobin ≥90 g/L.

Platelet count ≥100 × 10^9/L.

Total bilirubin <1.5 × ULN (upper limit of normal).

Creatinine <1.5 × ULN.

AST/ALT <1.5 × ULN.

Cardiac function: Left ventricular ejection fraction (LVEF) ≥55% by echocardiography.

Reproductive status: Women of childbearing potential must have a negative serum pregnancy test within 14 days prior to randomization.

ECOG performance status: ≤1.

Informed consent: Signed written informed consent.

3.2 Exclusion Criteria

Patients meeting any of the following criteria will be excluded:

Evidence of metastatic breast cancer:

Chest/abdominal CT and bone scan required at any time from diagnosis to randomization to exclude metastasis.

PET/CT may substitute for other imaging modalities.

Prior systemic therapy: Chemotherapy, endocrine therapy, targeted therapy, or radiotherapy for the current breast cancer.

Second primary malignancy, except:

Adequately treated non-melanoma skin cancer.

Prior immunotherapy: Treatment with anti-PD-1, anti-PD-L1, anti-PD-L2, or other immune checkpoint inhibitors.

Immune-related conditions:

Diagnosed immunodeficiency or active autoimmune disease.

Severe cardiopulmonary disease: Uncontrolled or clinically significant.

Active hepatitis: Hepatitis B or C with detectable viral load.

Transplant history: Prior organ or bone marrow transplantation.

Pregnancy or lactation: Pregnant or breastfeeding women.

Other contraindications: Severe uncontrolled comorbidities deemed by investigators to contraindicate chemotherapy or PD-1 inhibitor therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 357 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2030-03-31 (Estimated)

PRIMARY OUTCOMES:
PCR rate | At the time of surgery
  Total pathological complete response
PCR rate in PDL1 positive subgroup | At the time of surgery
  Total pathological complete response

SECONDARY OUTCOMES:
EFS | 5-10 years
  • Event-free survival (EFS)
DFS | 5-10 years
  Disease-free survival (DFS)
adverse events | up to 1 year
  Evaluate the nature, incidence and severity of chemotherapy adverse events according to CTCAE 5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Henan cancer hospital, Zhengzhou, Henan, China